CLINICAL TRIAL: NCT03319459
Title: FATE-NK100 as Monotherapy and in Combination With Monoclonal Antibody in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK-101
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: HER2 Positive Gastric Cancer; Colorectal Cancer; Head and Neck Squamous Cell Carcinoma; EGFR Positive Solid Tumor; Advanced Solid Tumors; HER2-positive Breast Cancer; Hepatocellular Carcinoma; Non Small Cell Lung Cancer; Renal Cell Carcinoma; Pancreatic Cancer; Melanoma
Keywords: Solid Tumor; HER2; EGFR; Advanced Solid Tumor; Breast Cancer; Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Colorectal Cancer; Gastric Cancer; HER2 Positive; EGFR Positive; EGFR+; HER2+; Immunotherapy; NK cell therapy; Natural killer cell therapy; antibody-dependent cell-mediated cytotoxicity; ADCC; Non small cell lung cancer; Renal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Pancreatic Neoplasms; Melanoma; Breast Neoplasms; Head and Neck Neoplasms; Stomach Neoplasms; Kidney Neoplasms | interventions — Cetuximab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Regimen A (Experimental): FATE-NK100 as a monotherapy in subjects with advanced solid tumor malignancies.
  Interventions: Drug: FATE-NK100
- Regimen B (Experimental): FATE-NK100 in combination with trastuzumab in subjects with human epidermal growth factor receptor 2 positive (HER2+) advanced breast cancer, HER2+ advanced gastric cancer or other advanced HER2+ solid tumors.
  Interventions: Drug: FATE-NK100; Drug: Trastuzumab
- Regimen C (Experimental): Regimen C: FATE-NK100 in combination with cetuximab in subjects with advanced colorectal cancer (CRC) or head and neck squamous cell cancer (HNSCC), or other epidermal growth factor receptor 1 positive (EGFR1+) advanced solid tumors.
  Interventions: Drug: FATE-NK100; Drug: Cetuximab

INTERVENTIONS:
Drug: FATE-NK100 — FATE-NK100 is a donor-derived NK cell product comprised of ex vivo activated effector cells with enhanced anti-tumor activity
Drug: Cetuximab — Epidermal growth factor receptor inhibitor antineoplastic agent
  Other Names: Erbitux
  Arms: Regimen C
Drug: Trastuzumab — HER2/neu receptor inhibitor
  Other Names: Herceptin
  Arms: Regimen B

SUMMARY:
This is a Phase 1, single-dose, open-label, dose-escalation study. The study will be conducted in three parts (i.e. regimens) in an outpatient setting as follows:

* Regimen A: FATE-NK100 as a monotherapy in subjects with advanced solid tumor malignancies.
* Regimen B: FATE-NK100 in combination with trastuzumab in subjects with human epidermal growth factor receptor 2 positive (HER2+) advanced breast cancer, HER2+ advanced gastric cancer or other advanced HER2+ solid tumors.
* Regimen C: FATE-NK100 in combination with cetuximab in subjects with advanced colorectal cancer (CRC) or head and neck squamous cell cancer (HNSCC), or other epidermal growth factor receptor 1 positive (EGFR1+) advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Regimen A only (monotherapy): Subjects with advanced metastatic solid tumors
2. Regimen B only (combination with trastuzumab): Subjects with advanced metastatic HER2+ solid tumors
3. Regimen C only (combination with cetuximab): Subjects with advanced metastatic EGFR+ solid tumors
4. Available related donor who is CMV+ and HLA-haploidentical or better but not fully HLA-matched
5. Presence of measurable disease by RECIST 1.1
6. Life expectancy of at least 3 months.
7. Provision of signed and dated informed consent form (ICF).
8. Stated willingness to comply with study procedures and duration.

Exclusion Criteria:

1. Females of reproductive potential that are pregnant or lactating, and males or females not willing to use a highly effective form of contraception from Screening through the end of the study.
2. Eastern Cooperative Oncology Group (ECOG) performance status >2.
3. Evidence of insufficient organ function as determined by the protocol.
4. Receipt of any biological therapy, chemotherapy, or radiation within 1 week of the Screening Visit and at least 3 weeks prior to Day 1, except for patients receiving maintenance trastuzumab.
5. Have central nervous system disease (CNS) as follows:

   1. Dose Escalation Cohorts: Active CNS disease, including history of CNS metastases.
   2. MTD/MFD Expansion Cohorts: CNS disease, including history of CNS metastases, that was not stable during the last 6 months.
6. Myocardial infarction (MI) within 6 months of Screening Visit.
7. Severe asthma.
8. Currently receiving or likely to require systemic immunosuppressive therapy from Day -7 to Day 29.
9. Uncontrolled infections.
10. Presence of any medical or social issues that are likely to interfere with study conduct, or may cause increased risk to subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | 28 days
  The incidence of dose-limiting toxicity (DLT) within each dose cohort within the first 28 days after FATE-NK100 administration (ie, Day 1 through Day 29).

SECONDARY OUTCOMES:
Objective-response rate (ORR) | 28 days, 57 days, 113 days, 169 days, 225 days, 281 days, 337 days, and 366 days.
  Objective-response rate (ORR): defined as the proportion of patients who achieve partial response (PR) or complete response (CR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at any time on study.
Pharmacokinetics (PK) of FATE-NK100 | 0 days, 1 day, 3 days, 5 days, 8 days, 12 days, 15 days, 22 days, 29 days, 43 days, 57 days, 85 days, 113 days
  The PK of FATE-NK100, as assessed by the proportion of lymphocytes in peripheral blood that are of donor/product origin at the specified time points.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Chou, MD, Study Director — Fate Therapeutics
Locations (4):
- United States (4):
  - UCSD Moores Cancer Center, San Diego, California
  - University of Minnesota, Minneapolis, Minnesota
  - The Ohio State University James Cancer Hospital, Columbus, Ohio
  - Baylor Scott & White Research Institute, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cichocki F, Valamehr B, Bjordahl R, Zhang B, Rezner B, Rogers P, Gaidarova S, Moreno S, Tuininga K, Dougherty P, McCullar V, Howard P, Sarhan D, Taras E, Schlums H, Abbot S, Shoemaker D, Bryceson YT, Blazar BR, Wolchko S, Cooley S, Miller JS. GSK3 Inhibition Drives Maturation of NK Cells and Enhances Their Antitumor Activity. Cancer Res. 2017 Oct 15;77(20):5664-5675. doi: 10.1158/0008-5472.CAN-17-0799. Epub 2017 Aug 8. PMID 28790065
- See also: GSK 3 inhibition drives maturation of NK cells and enhances their antitumor activity — https://www.ncbi.nlm.nih.gov/pubmed/28790065